CLINICAL TRIAL: NCT00595621
Title: Multi-Channel Gastric Electrical Stimulation for the Treatment of Gastroparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: GI Stimulation, Inc. (Industry); National Institutes of Health (NIH) (NIH); American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 9459
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Gastric Stasis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MGP-1 ON (Active Comparator): Experimental Pacemaker on for 6 weeks
  Interventions: Device: Enterra Multi-Channel Phased Gastric Pacemaker (MGP-1)
- MGP-1 OFF (Active Comparator): Experimental Pacemaker on or off for 4 weeks
  Interventions: Device: Enterra Multi-Channel Phased Gastric Pacemaker (MGP-1)

INTERVENTIONS:
Device: Enterra Multi-Channel Phased Gastric Pacemaker (MGP-1) — Multi-Channel Phased Gastric Pacemaker (MGP-1)

SUMMARY:
Investigate the safety and efficacy of multi-channel gastric electrical stimulation in the treatment of patients with severe diabetic gastroparesis refractory to standard therapy.

DETAILED DESCRIPTION:
Evaluation of severe symptom control of nausea, vomiting, postprandial fullness, early satiety, bloating and discomfort related to drug refractory gastroparesis present as a GI complication in diabetic patients. External gastric pacemaker system will be placed at the same time of implantation of Enterra (internal gastric stimulator-permanent device) to assess symptoms, quality of life improvement and investigate the changes in gastric emptying time in diabetic gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

* Severe nausea and vomiting for at least 6 months
* Documented delayed gastric emptying
* Failed extensive medical treatment

Exclusion Criteria:

* Previous gastric surgery
* Pregnancy or planned pregnancy
* Primary eating or swallowing disorders
* Scheduled or planned MRI testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W. McCallum, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Diabetic gastroparetic patients who qualified to participate in this study based on inclusionary criteria were recruited from the Gastroenterology Motility Clinic of KUMC in Kansas City, KS
Pre-assignment Details: All subjects underwent an open-label phase where multi-channel gastric pacemaker (MGP-1) was turned "ON" for 6 weeks. After this phase they were randomized in double blind fashion to MGP-1 "ON" or "OFF" for another 4 weeks. 3 participants were not randomized to continue the study after the open-label phase.
Groups:
- MGP-1 "ON": Experimental Pacemaker on for 6 weeks during the open label phase then on for 4 weeks during the randomization phase.
  Enterra Multi-Channel Phased Gastric Pacemaker (MGP-1): Multi-Channel Phased Gastric Pacemaker (MGP-1)
- MGP-1 "OFF": Experimental Pacemaker on for 6 weeks during the open label phase then off for 4 weeks during the randomization phase.
  Enterra Multi-Channel Phased Gastric Pacemaker (MGP-1): Multi-Channel Phased Gastric Pacemaker (MGP-1)
Period: Open Label Run in
Arm/Group | MGP-1 "ON" | MGP-1 "OFF"
Started | 22 | 0
Completed | 19 | 0
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Randomization and Study
Arm/Group | MGP-1 "ON" | MGP-1 "OFF"
Started | 10 | 9
Completed | 8 | 8
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MGP-1 "ON" | MGP-1 "OFF" | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 42 [27 to 58] | 40 [31 to 60] | 42 [27 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Slow Wave Entrainment
Description: Participants were monitored for up to 3 months. Measure is the percent of normal slow waves (2-4 cpm) generated by MGP-1 device while it was ON or OFF
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: percentage of slow waves entrainment
Arm/Group | MGP-1 "ON" | MGP-1 "OFF"
Number analyzed (Participants) | 8 | 8
percentage of slow waves entrainment
  Baseline Pre-Randomization Phase | 72 (3) | 70 (2)
  Post-Randomization Phase | 84 (2) | 78 (1.5)

2. Secondary Outcome: The Percent (Percentage) of Gastric Retention of a Solid Meal
Description: The retention of a study meal was measured at baseline, 1,2,3 and 4 hours of the test. The percent of food retained in a stomach at 4 hours was compared when MGP-1 was ON and OFF.
Time Frame: 12 Weeks
Measure: Number; unit: percent of food retained
Arm/Group | MGP-1 "ON" | MGP-1 "OFF"
Number analyzed (Participants) | 8 | 8
percent of food retained
  Baseline Pre-Randomization Phase | 46 | 36
  Post-Randomization Phase | 33 | 42

3. Secondary Outcome: Severity of Gastroparetic Symptoms
Description: Measure represents change in symptom severity as measured by a self assessment Symptom Interview Form evaluating severity of vomiting, nausea, early satiety, bloating, postprandial fullness, epigastric pain, and epigastric burning. Symptoms were rated from 0 - absence of symptom to 4 - extremely severe. The overall score was calculated from the sum of seven symptom sub-scores with a total possible score range of 0 - absence of all symptoms to 28 - all symptoms extremely severe.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MGP-1 "ON" | MGP-1 "OFF"
Number analyzed (Participants) | 8 | 8
units on a scale
  Baseline Pre-Randomization Phase | 13 (1.2) | 14 (1)
  Post-Randomization Phase | 6 (1.1) | 16 (1.1)

4. Secondary Outcome: Changes in Quality of Life (QoL) Assessment (Physical (P) and Mental (M))
Description: Measure represents percentage change from baseline to end of study. QoL measured using the Short Form Health Survey (SF-36) questionnaire. The SF-36 is a generic measure of QoL. Physical QoL (Physical Component Summary; PCS) and emotional QoL (Mental Component summary; MCS) scale components of the survey used for outcome. Scores range from 0 to 100 with lower scores indicating more disability and higher scores less disability.
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: percentage change in scale score
Arm/Group | MGP-1 "ON" | MGP-1 "OFF"
Number analyzed (Participants) | 8 | 8
percentage change in scale score
  Physical Score | 60 (21) | 30 (11)
  Mental Score | 55 (19) | 40 (14)

5. Secondary Outcome: Changes in Hemoglobin A1c (HbA1c) Level
Description: HbA1c was evaluated at the baseline and after completion of all the phases of the study
Time Frame: 12 Weeks
Measure: Mean (Full Range); unit: % HbA1c
Arm/Group | MGP-1 "ON" | MGP-1 "OFF"
Number analyzed (Participants) | 8 | 8
% HbA1c | 8.1 [7.6 to 10.3] | 8.2 [8.0 to 11.0]

6. Secondary Outcome: Changes in Hospital Admissions
Description: Measured by days of hospitalization per patient. Number of days of hospitalization was recorded at baseline and after completion of all phases of the study.
Time Frame: 12 Weeks
Measure: Mean (Full Range); unit: days
Arm/Group | MGP-1 "ON" | MGP-1 "OFF"
Number analyzed (Participants) | 8 | 8
days | 1.5 [0 to 4] | 2.1 [0 to 7]

ADVERSE EVENTS:
Time Frame: Duration of the study, up to 12 weeks.
Groups:
- Open Label Run: Experimental Pacemaker on for 6 weeks during the open label phase (preceding MGP-1 "ON" and MPG-1 "OFF" randomization phases).
  Enterra Multi-Channel Phased Gastric Pacemaker (MGP-1): Multi-Channel Phased Gastric Pacemaker (MGP-1)
- MPG-1 "OFF": Experimental Pacemaker on for 6 weeks during the open label phase then off for 4 weeks during the randomization phase.
  Enterra Multi-Channel Phased Gastric Pacemaker (MGP-1): Multi-Channel Phased Gastric Pacemaker (MGP-1)
Arm/Group | Open Label Run | MGP-1 "ON" | MPG-1 "OFF"
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 1/22 | 2/10 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Run (N=22) | MGP-1 "ON" (N=10) | MPG-1 "OFF" (N=9)
Dislodgement of the electrode(s) (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Technical issue with the MGP-1 system (Product Issues) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes